CLINICAL TRIAL: NCT07119294
Title: Molecular Imaging of Cancer-associated Fibroblasts in Glioblastoma: a FAPI PET/MR Study.
Acronym: GlioFAPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IJB-NM-GlioFAPI
Record Dates: First submitted 2025-07-15; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma
Keywords: glioblastoma; FAPI PET/CT
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: * Patients with a brain lesion suspected of glioblastoma based on imaging will receive a FAPI PET-MR before surgery, matched with the usual examinations (MRI and FET PET-CT).
  * Patients with suspected glioblastoma recurrence in their follow-up: a FAPI PET/MR, matched with the usual examinations (MRI and FET PET-CT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with a brain lesion suspected of glioblastoma based on imaging with a FAPI PET-MR before s (Other)
  Interventions: Diagnostic Test: FAPI PET/MR
- patients with suspected glioblastoma recurrence in their follow-up. (Other)
  Interventions: Diagnostic Test: FAPI PET/MR

INTERVENTIONS:
Diagnostic Test: FAPI PET/MR — FAPI PET/MR prior surgery or during recurrence suspiscion

SUMMARY:
Glioblastoma is a highly aggressive and malignant form of brain cancer that arises from the glial cells of the brain. It is the most common and deadliest type of primary brain tumor in adults, with a very poor prognosis and a low survival rate. Glioblastoma is characterized by rapid and uncontrolled growth, infiltrative invasion into surrounding brain tissue, and resistance to standard treatments. Therefore, new therapeutic strategies are highly needed. A subpopulation of fibroblasts called "cancer-associated fibroblasts" (CAFs) is know to be a key constituent of tumor stroma in several non-CNS tumors (e.g., breast, colon, lung,ovarian, or pancreatic cancers) . These CAFs express a specific protein called "fibroblast activation protein" (FAP), which is usually not expressed in healthy adult mammalian tissues. FAP has been shown to be elevated in vitro and in situ in glioblastoma cells , suggesting that CAFs expressing FAP might also play a functional role in malignant brain tumors. This research project aims at better characterizing the links between areas of increased FAPI uptake within glioblastomas and the local level of tumor aggressiveness. This will be done by comparing the distribution of their anatomical locations uptake within the tumor with the distribution of the uptake of other markers of local tumor aggressiveness such as amino-acid PET (FET), and MRI measures of cerebral blood flow such as arterial spin labelling (ASL) or perfusion-weighted echo-planar images . Ultimately, when possible, neuroimaging data will be compared with pathology findings from targeted brain biopsy samples or material from ablative surgery. Furthermore, this study will provide the necessary first step towards more large scale studies evaluating the potential use of 177Lu-FAPI as therapeutic agent in glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Age above or equal to 18 years
* Patients with a brain lesion suspected of glioblastoma based on neuroimaging data or patients with suspected recurrence of glioblastoma
* ECOG performance status ≤ 3
* Signed Informed Consent form (ICF) obtained prior to any study related procedure.

Exclusion Criteria:

* Pregnant and/or lactating women.
* Subject with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.
* Claustrophobic patient
* Known hypersensitivity reactions to the FAPI or to any excipients, or to gadolinium-based contrast agents (GBCAs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
To compare the FAPI uptake within the tumor using quantitative measures (SUVmax, SUVmean, and volume) with the uptake of other markers of local tumor aggressiveness such as amino-acid PET and MRI data. | up to 4 weeks : from enrollment until surgery date or the end of recurrence follow up
To compare FAPI tumor uptake (SUVmax, SUVmean) with FAP expression based on anatomopathological analysis (Immunohistochemistry) from targeted brain biopsy samples or material from ablative surgery | up to 4 weeks : from enrollment until anapathological analysis

SECONDARY OUTCOMES:
To compare FAPI uptake (SUVmax, SUVmean, Volume) and amino-acid PET uptake in case of tumor recurrence and in case of radionecrosis | up to 4 weeks : from enrollment to FET PET exam date

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium